CLINICAL TRIAL: NCT03678857
Title: The Effect of Creatine Timing on Resistance Training Adaptations: A Within-subject Design
Brief Title: Creatine Timing and Resistance Training Adaptations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22261
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: creatine, hypertrophy, strength
MeSH Terms: conditions — Hypertrophy | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An independent researcher will label the placebo and creatine and only reveal which group is which after data has been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Before (Experimental): Receives Creatine before and placebo after training.
  Interventions: Dietary Supplement: Creatine
- Creatine After (Experimental): Receives creatine after and placebo before training.
  Interventions: Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: Creatine — Participants will resistance train their left arm and left leg one day and their right arm and right leg the next day. Participants will supplement with creatine BEFORE one of the training days (randomized to either left or right side) and on the opposite training day (opposite side of the body to the previous training day) supplement with creatine AFTER training. Having the same person in both conditions will control for genetics, habitual diet, other daily activities, and so on, that may have confounded previous research. Muscle mass and strength changes will be measured in each limb prior to and following 8 weeks of training to determine whether creatine timing influenced muscle growth.
  Research Question: To determine whether creatine supplementation timing (i.e., before versus after training) effects 8 weeks of resistance training adaptations (i.e., muscle growth and strength changes).

SUMMARY:
Emerging evidence suggests that the timing of creatine supplementation may be an important regulator of muscle growth and strength. It is unclear whether creatine ingested before or after resistance training is more beneficial. A limitation of previous research is the use of a between subject design. A between subject design is associated with several potential confounders (habitual diet, genetics, activities of daily living, etc.) that may have masked the true effect. The purpose of this study is to examine the effect of creatine timing (creatine before vs. creatine after) using a randomized, double blind, repeated measures, within-subject design. Participants will resistance train their left arm and left leg one day and their right arm and right leg the next day. Participants will supplement with creatine BEFORE one of the training days (randomized to either left or right side) and on the opposite training day (opposite side of the body to the previous training day) supplement with creatine AFTER training. Having the same person in both conditions will control for genetics, habitual diet, other daily activities, and so on, that may have confounded previous research. Muscle mass and strength changes will be measured in each limb prior to and following 8 weeks of training to determine whether creatine timing influenced muscle growth.

Research Question: To determine whether creatine supplementation timing (i.e., before versus after training) effects 8 weeks of resistance training adaptations (i.e., muscle growth and strength changes).

DETAILED DESCRIPTION:
Emerging evidence suggests that the timing of creatine supplementation may be an important regulator of muscle growth and strength. It is unclear whether creatine ingested before or after resistance training is more beneficial. A limitation of previous research is the use of a between subject design. A between subject design is associated with several potential confounders (habitual diet, genetics, activities of daily living, etc.) that may have masked the true effect. The purpose of this study is to examine the effect of creatine timing (creatine before vs. creatine after) using a randomized, double blind, repeated measures, within-subject design. Participants will resistance train their left arm and left leg one day and their right arm and right leg the next day. Participants will supplement with creatine BEFORE one of the training days (randomized to either left or right side) and on the opposite training day (opposite side of the body to the previous training day) supplement with creatine AFTER training. Having the same person in both conditions will control for genetics, habitual diet, other daily activities, and so on, that may have confounded previous research. Muscle mass and strength changes will be measured in each limb prior to and following 8 weeks of training to determine whether creatine timing influenced muscle growth.

Methods:

Day 1 - A 3-day dietary record (to determine typical energy intake and macronutrient breakdown for participant characteristics), anthropometric testing (height and weight), age, muscle thickness (via ultrasound for elbow flexors and leg extensors), and bicep curl and leg extension 1-repetition maximal strength will be determined. In addition, strength training experience and hand dominance will be determined via standardized questionnaires. Muscle thickness of the elbow flexors and leg extensors will be measured before and after the 8 weeks training period using B-mode ultrasound (LOGIQ e BTO8, GE Healthcare, Milwaukee, Wisconsin, USA). Bicep curl and leg extension maximal strength will be assessed on each limb using a 1-repetition maximum (1-RM) standard testing procedure. Briefly, following 5 minutes of cycling on a stationary cycle ergometer, participants will perform 2 warm-up sets (to reduce the risk of injury) in the following order: 1 set of 10 repetitions using a weight determined by each subject to be comfortable and 1 set of 5 repetitions using increased weight. Two minutes after the warm-up sets, weight will be progressively increased for each subsequent 1-repetition maximum attempt with a 2-min rest interval. The 1-rep max will be reached in 4-6 sets, excluding the 2 warm-up sets. All exercise testing will be superivsed by a a trained research assistant or by a Canadian Society for Exericse Physiology certified exercise physiologist.

Next 8 Weeks (Resistance Training Program):

The Resistance Training will include 3 to 6 sets (progressing overtime; starting at 3 sets and increasing 1 set per week until a maximum of 6 sets) of 80% of 1 repetition maximum with a 3 second eccentric phase (i.e., 1-2 seconds up and 3 seconds down) until failure (unable to complete another repetition or form failure). Each participant will complete 3 training sessions per week per side (total of 6 sessions per week). Prior to each training session, but after the supplement had been consumed, each participant will perform a 5-min stationary cycling warm-up at a self-selected intensity. Resistance exercises will include bicep curls and leg extensions. These two exercises were selected because they are safe and easy to learn and include large upper body and lower body musculature that are known to respond to resistance training. Participants will maintain daily training logs that include the weight, number of sets, and number of repetitions.

Supplementation Protocol:

Participants will supplement with creatine on one of the training days (either when they are training their left or right side) BEFORE training in a dose previous shown to enhance training adaptations (0.1 grams of creatine per kilogram of body weight before training and a placebo - cornstarch maltodextrin after training). When the participants trains their opposite side of the body they will supplement with creatine AFTER training (0.1 grams per kilogram of placebo before and 0.1 grams per kilogram of creatine after). The placebo will be identical in color, texture, tast, and appearance. The purpose of the placebo is so the participants will not know which day they are receiving creatine before training and which day they are receiving creatine after training. The creatine is research grade and has been independtly tested and will be provided free of charge. Any adverse events related to the exercise or the supplement will be recorded.

Post Testing:

Following the 8 weeks of training. Participants will complete the baseline testing (Day 1) protocols to determine strength and muscle thickness changes in each limb.

ELIGIBILITY:
Inclusion Criteria:

* You may be able to participate in this study if you are between the ages of 18 and 35, are free of disease (e.g., diabetes), do not currently take creatine or other supplements (within the last 12 weeks), and have no known cardiovascular disease or other medical conditions which prevent you from performing physical activity or this type of nutritional supplement.

You must also have no other reasons that might make exercise unsafe for you. You will complete a questionnaire (Get Active Questionnaire) to help identify any illness or health concern that could be worsened by performing exercise or make exercise unsafe for you.

Exclusion Criteria:

* You will not be eligible to participate in this study:

  1. If your doctor has informed you that you have a heart condition and should only do physical activity recommended by a doctor.
  2. If you feel pain in your chest when you perform any physical activity.
  3. If in the past the month you have had chest pain when you were not doing any physical activity.
  4. If you lose your balance or consciousness because of dizziness.
  5. If you have bone or joint problem (for example, back, knee, or hip) that could be made worse by a change in your physical activity.
  6. You have previously had a heart attack or stroke
  7. If you know of any other reason why you should not do physical activity.
  8. You currently take creatine supplements and/or other "performance enhancing" nutritional supplements

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Hypertrophy (Muscle thickness will be determined via ultrasound) | 8 weeks
  Muscle thickness will be determined via ultrasound.
Strength (1 repetition maximum will be determined via standard 1RM protocols) | 8 weeks
  1 repetition maximum will be determined via standard 1RM protocols

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Forbes, PhD, Principal Investigator — Brandon University
Locations (1):
- Brandon University, Brandon, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No